CLINICAL TRIAL: NCT00885729
Title: Mesenchymal Stem Cells in a Clinical Trial to Heal Articular Cartilage Defects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, MD, PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-0738c 2009
Record Dates: First submitted 2009-04-17; First posted 2009-04-22 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Defect of Articular Cartilage
Keywords: Cartilage defect; chondrocytes; mesenchymal stem cells (MSC); femoral condyle; knee
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem cells (Experimental): Cartilage defect are treated surgical either with chondrocytes or stem cells
  Interventions: Procedure: stem cells; Procedure: Chondrocytes
- Rehabilitation (Active Comparator): Active rehabilitation program
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Procedure: stem cells — Stem cells or chondrocytes under a commercial available membrane
  Arms: Stem cells
Procedure: Chondrocytes — Implantation of chondrocytes
  Arms: Stem cells
Other: Rehabilitation program — Strength exercises, neuromuscular exercises
  Arms: Rehabilitation

SUMMARY:
The purpose of this study is to:

* Compare the treatment efficacy of autologous mesenchymal stem cells (Mesenchymal Stem Cells) versus chondrocytes implanted in a commercial available scaffold in a human clinical trial.
* Determine the effects of specific three months strength training program preoperatively to improve knee function and possible postpone the need of cartilage repair surgery.
* Determine if degenerative changes occur in the knee joints following cartilage repair. This question will be investigated in the proposed clinical trial.
* Determine the characteristics of patients treated either by surgery or by rehabilitation in a long-term follow-up (1, 5 years).

DETAILED DESCRIPTION:
Musculoskeletal diseases are growing in the Norwegian population and are currently the largest group of the chronic diseases (31%). Musculoskeletal diseases are the largest cause of disability on the working part of our population (49%). The most frequent problems are rheumatism, osteoarthritis and unspecific back pain. The most common known etiology is traumatic events towards the joint. Often, the degenerative development starts with a small injury to the cartilage on weightbearing surface of the joint. This leads to changes in the surrounding cartilage, indicative of degenerative joint disease or arthrosis. When the injured area becomes larger than 2 cm2, the patients seem to experience pain. Our group has shown that 11% of patients, who underwent an arthroscopy for knee pain, had a cartilage injury on weightbearing surface with depth down to bone (grade IV) (Aroen et al.).Unfortunately, articular cartilage shows a very limited capacity of healing. Several surgical techniques have been developed to fill the cartilage defects, but so far none of them have been able to produce normal cartilage Chondrocyte implantation techniques are at date the most popular treatment, but have not demonstrated their superiority to other cartilage repair techniques. Some clinical randomised studies exist though a more thorough review of the cartilage repair methods in a study by Jakobsen and coauthors verified that no conclusion could be made considering treatment options for articular cartilage injury (Jakobsen, Engebretsen, and Slauterbeck). Although the natural history of these lesions is not finally outlined it is clear that for some patients the disruption of the cartilage surface imposes disability especially for the young athlete. The clinical studies report a significant improvement from the preoperative status although full knee function is not obtained with either of the techniques available today (Bentley et al.;Brittberg et al.;Horas et al.;Knutsen et al.). The expected Lysholm score of 80 and the standard deviation tends to be large or is not reported which illustrating the considerable variation and that full knee function is not obtained (Peterson et al.).The impact of disrupting the cartilage surface to obtain chondrocytes for culturing has not gained much attention in the clinical studies using this repair method. However it is reported that adverse effects exist as a result of this harvesting of chondrocytes for culturing (Whittaker et al.). Whittaker and coauthors observed that the harvesting of chondrocytes for cell culturing and subsequent implantation in talus resulted in a mean 15 points reduction in Lysholm score in 7 out of 10 patients. Furthermore, additional even in the best hands a mean Lysholm score of 79 are obtained for a single lesion at the femoral condyle (Peterson et al.). Even though the new scaffolds seem to reduce the rate of reoperation as a result of graft hypertrophy from 21 % to 9 %, the harvesting procedure of cartilage may still contribute to the suboptimal by this approach (Bartlett et al.;Gooding et al.). Consequently, there is a need for a better causing less morbidity when harvesting. Mesenchymal stem cells (MSC) represent an alternative cell source with the potential of generating hyaline cartilage without the same adverse effects. In addition with MSC more cells will be available for culturing with the potential of treatment of larger lesions possible. Furthermore, the repair potential of mesenchymal stem cells is not expected to decrease with age indicating that also the aging athlete may benefit from a procedure based on cartilage repair with this cell source (Dressler, Butler, and Boivin). The use of mesenchymal stem cell aspirate from the iliaca crest under a periosteum flap support the view that this might be an option to treat knee cartilage defects with success, although this study also has periosteum hypertrophy as a side effect in one of the patients (Slynarski, Deszczynski, and Karpinski). The beneficial effects of this therapy has also been reported in other studies both clinical and experimental ones (Takagi et al.;Wakitani et al.;Wakitani et al.;Wakitani et al.). Thus, the current project will investigate if the similar results can be obtained with mesenchymal stem cells as with chondrocytes both delivered in a commercial available scaffold in clinical trial with patients eligible for the current treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian citizens
* A full-thickness cartilage lesion (diameter > 15 mm, but less than 6 cm2 and Lysholm score < 75 points) located on the femoral condyle

Exclusion Criteria:

* Patients with malignment of the knee
* Other knee pathology such as ACL injury or a nontreated meniscus injury will not be included in the study to avoid the impact of these knee pathologies on the final results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Lysholm score | 2018

SECONDARY OUTCOMES:
Radiographics | Two and five years

OTHER OUTCOMES:
Return to work | 1 Year
  Return to work one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lars Engebretsen, MD,PhD, Study Chair — Professor
Locations (1):
- Oslo UniversityHospital-Ullevaal, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Aroen A, Brogger H, Rotterud JH, Sivertsen EA, Engebretsen L, Risberg MA. Evaluation of focal cartilage lesions of the knee using MRI T2 mapping and delayed Gadolinium Enhanced MRI of Cartilage (dGEMRIC). BMC Musculoskelet Disord. 2016 Feb 11;17:73. doi: 10.1186/s12891-016-0941-y. PMID 26868015
- [Derived] Rotterud JH, Reinholt FP, Beckstrom KJ, Risberg MA, Aroen A. Relationship between CTX-II and patient characteristics, patient-reported outcome, muscle strength, and rehabilitation in patients with a focal cartilage lesion of the knee: a prospective exploratory cohort study of 48 patients. BMC Musculoskelet Disord. 2014 Mar 24;15:99. doi: 10.1186/1471-2474-15-99. PMID 24661577
- [Derived] Wondrasch B, Aroen A, Rotterud JH, Hoysveen T, Bolstad K, Risberg MA. The feasibility of a 3-month active rehabilitation program for patients with knee full-thickness articular cartilage lesions: the Oslo Cartilage Active Rehabilitation and Education Study. J Orthop Sports Phys Ther. 2013 May;43(5):310-24. doi: 10.2519/jospt.2013.4354. Epub 2013 Mar 13. PMID 23485794